CLINICAL TRIAL: NCT07254416
Title: To Evaluate the Efficacy and Safety of NEPA Combined With Megestrol Acetate Versus NEPA Combined With Dexamethasone in Preventing Nausea and Vomiting Caused by T-DXd in Breast Cancer Patients
Brief Title: A Study on Nausea and Vomiting Caused by T-DXd in Breast Cancer Patients
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Collaborators: Shaanxi Provincial Cancer Hospital (Other); The First Affiliated Hospital of Henan University of Science & Technology (Unknown); Shanxi Bethune Hospital (Other); Tianjin Cancer Hospital Airport Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AKZ-ADC-01
Record Dates: First submitted 2025-11-19; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer Patients Treated With T-DXd
Keywords: NEPA; Netupitant and Palonosetron Hydrochloride Capsules; megeprogesterone acetate; dexamethasone
MeSH Terms: interventions — Dexamethasone; Megestrol Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NEPA+ Megestrol Acetate (Experimental)
  Interventions: Drug: NEPA; Drug: Megestrol Acetate
- NEPA+ Dexamethasone (Active Comparator)
  Interventions: Drug: NEPA; Drug: Dexamethasone

INTERVENTIONS:
Drug: NEPA — On the first day, oral administration of NEPA(netopitan 300mg+ palonosetron 0.50mg)
Drug: Dexamethasone — On the first day, oral administration of dexamethasone 6mg; From the 2nd to the 4th day, take dexamethasone 3.75mg orally per day.
  Arms: NEPA+ Dexamethasone
Drug: Megestrol Acetate — From the 1st to the 10th day, take 160mg of Megestrol Acetate orally per day.
  Arms: NEPA+ Megestrol Acetate

SUMMARY:
This study was a multicenter, prospective, controlled trial involving 120 breast cancer patients receiving T-DXd-based therapy. Participants were randomly assigned to either the experimental group (NEPA plus megestrol acetate) or the control group (NEPA plus dexamethasone), with 60 patients in each group. The intervention was administered over two treatment cycles. During this period, the onset time, frequency, and severity of nausea and vomiting were recorded and subjected to statistical analysis.

The primary objective of this study was to evaluate the efficacy and safety of netupitant/palonosetron capsules (NEPA) combined with megestrol acetate compared to the standard triple antiemetic regimen (NEPA plus dexamethasone) in preventing chemotherapy-induced nausea and vomiting (CINV) in breast cancer patients undergoing T-DXd-containing regimens. The findings aim to generate clinical evidence to support optimal antiemetic management, minimize the risk of dose reduction or treatment discontinuation due to gastrointestinal adverse events, and ultimately improve patient quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. The patient is at least 18 years of age;
2. The patient has a histologically or cytologically confirmed diagnosis of breast cancer;
3. The patient is receiving full-dose trastuzumab deruxtecan (T-DXd) monoclonal antibody therapy for the first time;
4. The patient has an Eastern Cooperative Oncology Group (ECOG) performance status score of 2 or lower;
5. The patient voluntarily agrees to comply fully with the study protocol requirements and has provided written informed consent.

Exclusion Criteria:

1. The patient is currently taking medications that may interfere with the assessment of nausea or vomiting, including but not limited to other 5-HT3 receptor antagonists, NK1 receptor antagonists, psychotropic agents, or opioid analgesics;
2. The investigator determines that the patient's nausea or vomiting is highly likely attributable to anti-tumor treatments not involving antibody-drug conjugate (ADC) therapy;
3. The patient is deemed unsuitable for glucocorticoid or progesterone use;
4. The patient has a history of hypersensitivity to netupitant, palonosetron, or any excipient in the capsule formulation;
5. The patient has significant gastrointestinal conditions affecting oral drug absorption, such as dysphagia, chronic diarrhea, or intestinal obstruction;
6. The patient has a severe psychiatric disorder or difficulties understanding the study procedures, completing questionnaires, or communicating effectively in Chinese;
7. The investigator identifies any other condition that may compromise the conduct of the clinical study or the interpretation of its results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
The CR rate within 0-120 hours (0-5 days) after the first cycle of T-Dxd treatment | 0-120 hours (0-5 days)

SECONDARY OUTCOMES:
The CR rates of 0-24 hours, 24-120 hours, 120-240 hours and 0-504 hours after the first and second cycles of T-Dxd treatment. | 0-24 hours, 24-120 hours, 120-240 hours and 0-504 hours
The CR rate within 0-120 hours (0-5 days) after the first cycle of T-Dxd treatment | 0-120 hours (0-5 days)
The CC rates of 0-24 hours, 24-120 hours, 0-120 hours, 120-240 hours and 0-504 hours after the first and second cycles of T-Dxd treatment. | 0-24 hours, 24-120 hours, 0-120 hours, 120-240 hours and 0-504 hours
The time and duration of the first significant nausea and vomiting. | From the administration of T-Dxd to 21 days
The proportion of patients undergoing salvage treatment. | From the administration of T-Dxd to 21 days
The incidence of ADC reduction due to adverse reactions | From the administration of T-Dxd to 21 days
Evaluation of the EORTC QLQ-C30 (version 3) Quality of Life Questionnaire. | From the administration of T-Dxd to 21 days

IPD SHARING:
Plan to Share IPD: No